CLINICAL TRIAL: NCT05454306
Title: The Anser Clavicle Pin for Surgical Management of Midshaft Clavicle Fractures; A U.S. Prospective Case Series
Brief Title: Anser Clavicle Pin for Surgical Management of Midshaft Clavicle Fractures
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: funding
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORSU-2022-31047
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Clavicle Fracture
Keywords: Clavicle fracture; Clavicle pin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Anser Clavicle Pin (Experimental): Patients treated with Anser Clavicle Pin in the setting of a displaced midshaft clavicle fracture
  Interventions: Device: Anser Clavicle Pin

INTERVENTIONS:
Device: Anser Clavicle Pin — The Anser Clavicle Pin is an intramedullary device that has been studied in 20 patients in an EU-based prospective case series.28 A 100% union rate was found. The Constant-Murley score at 1-year was 96.7 (SD 5). The Disabilities of Arm, Shoulder and Hand score was 5.1 (SD 10). There were no infections, neuropathy of the supraclavicular nerve or hardware irritation requiring removal of hardware. Three device-related complications (15%) occurred including plastic deformation, protrusion and hardware failure. VAS satisfaction was 8.9 (SD 1) at the 1-year follow up.

SUMMARY:
The goals of this multi-site study are to evaluate the union rate, patient satisfaction, and functional results of the Section 510(K) approved Anser Clavicle Pin in a prospective 50 patient clinical trial in a U.S. population.

ELIGIBILITY:
Inclusion Criteria:

* Displaced midshaft clavicle fracture Type 2B according to the Robinson Classification
* Skeletally mature
* Surgery performed within 4 weeks after trauma

Exclusion Criteria:

* Not fit for surgery by the anesthesiologist
* Nonunion or previous malunion
* Possible noncompliant patients (eg, alcohol and drug addiction, dementia)
* Additional neurovascular injury
* Pathologic fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2028-01-09 (Estimated); Primary Completion 2030-01-09 (Estimated); Study Completion 2030-01-09 (Estimated)

PRIMARY OUTCOMES:
ASES Score- 2 week | 2 weeks post-operation
  American Shoulder and Elbow Surgeons Score
ASES Score- 6 week | 6 weeks post-operation
  American Shoulder and Elbow Surgeons Score
ASES Score- 3 month | 3 months post-operation
  American Shoulder and Elbow Surgeons Score
ASES Score- 1 year | 1 year post-operation
  American Shoulder and Elbow Surgeons Score
DASH Score- 2 week | 2 weeks post-operation
  Disabilities of Arm, Shoulder and Hand Score
DASH Score- 6 week | 6 weeks post-operation
  Disabilities of Arm, Shoulder and Hand Score
DASH Score- 3 month | 3 months post-operation
  Disabilities of Arm, Shoulder and Hand Score
DASH Score- 1 year | 1 year post-operation
  Disabilities of Arm, Shoulder and Hand Score
Radiographic union rate | 1 year post-operation
  Radiographic union is defined as a 2/3rd circumferential cortical bridging between medial and lateral fragments on both radiographs as determined by the treating surgeon and an independent radiologist
Clinical union rate | 1 year post-operation
  Clinical union is defined as the absence of pain over the fracture site upon palpation.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Braman, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States